CLINICAL TRIAL: NCT01499108
Title: Time Course of the Blood Pressure Lowering Effect of Liraglutide Therapy in Type 2 Diabetes
Acronym: Liratime
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Peter Rossing (Other)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor-Investigator, Peter Rossing, Director of Research, Chief Physician, DMSc, Steno Diabetes Center Copenhagen
Organization: Steno Diabetes Center Copenhagen (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011-005344-95
Record Dates: First submitted 2011-12-12; First posted 2011-12-26 (Estimated); Last update posted 2015-02-02 (Estimated); Status verified 2013-07

CONDITIONS: Type 2 Diabetes
Keywords: type 2 diabetes; hypertension; liraglutide; kidney function
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypertension | interventions — Liraglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Liraglutide (Experimental): single-group study were participants recieve Liraglutide
  Interventions: Drug: liraglutide

INTERVENTIONS:
Drug: liraglutide — Subcutaneous injection of liraglutide at doses of 0.6, 1.2, and 1.8 mg once daily during the 49 days duration of the study
  Other Names: Victoza

SUMMARY:
Background: Preclinical blood pressure (BP) data from studies of hypoglycemic effects of liraglutide treatment (the LEAD program), revealed a significant antihypertensive potential. The time course and the mechanism behind this effect are unknown.

Objectives: To evaluate the time course of the antihypertensive effect of liraglutide treatment in patients with type 2 diabetes

Design: Open-label study with intervention and subsequent washout period

Patient Population: 35 hypertensive (SBP ≥130 mm Hg and DBP ≥80 mmHg) patients with type 2 diabetes.

Intervention: All patients will be treated with liraglutide 0.6 mg once daily for 7 days and will then be titrated to 1.2 mg once daily for 14 days and then titrated to 1.8 mg once daily for 4 weeks. This is followed by a washout period of 3 weeks without liraglutide treatment.

Endpoints: 24-hour blood pressure, natriuresis, extra cellular volume (ECV

DETAILED DESCRIPTION:
Hypotheses Primary hypothesis • Liraglutide treatment causes a reduction in 24h BP

Secondary hypothesis:

* The effect on BP may be mediated by an increase in natriuresis, thereby affecting ECV
* The effect on BP may be mediated by a decrease in arterial stiffness and central aortic pressure

Purpose Primary purpose

• To assess how quickly the antihypertensive effect of liraglutide treatment set in after initiation in patients with type 2 diabetes

Secondary objectives

* To measure the effect of liraglutide treatment on natriuresis.
* To measure the effect of liraglutide treatment on ECV
* To measure the effect of liraglutide treatment on arterial stiffness
* To measure weight change after initiation of liraglutide treatment

ELIGIBILITY:
Inclusion Criteria:

1. Must give written informed consent before participation. Patient information and consent form must be approved by the Danish Medicines Agency and the Regional Scientific Ethical Committee
2. Male or female patients > 18 years with type 2 diabetes (WHO criteria).
3. Patients must be on treatment with metformin. Any form of treatment with SU compounds will be discontinued and washed out for two weeks prior to the start of study drug.
4. eGFR ≥ 60 ml/min/1.73 m2 (estimated by MDRD formula)
5. Fertile female patients must use chemical, hormonal and mechanical contraceptives or be in menopause (i.e. must not have had regular menstrual bleeding for at least one year) or have undergone bilateral oophorectomy or have been surgically sterilized or hysterectomised at least six months prior to screening
6. Patients must be on antihypertensive treatment or having elevated blood pressure (SBP ≥130 mm Hg and DBP ≥80 mmHg), lower than 170/105 mm Hg at baseline and the patients must be stable antihypertensive medication for at least 4 weeks prior to baseline
7. Patients must be on stable hypoglycemic medication for at least two weeks before the first visit.
8. Must be able to communicate with the investigator

Exclusion Criteria:

1. Ongoing insulin therapy
2. BP > 170/105 mm Hg at baseline
3. Type 1 diabetes mellitus
4. Chronic pancreatitis / previous acute pancreatitis
5. Known or suspected hypersensitivity to trial product(s) or related products.
6. Treatment with oral glucocorticoids, calcineurin inhibitors, or dipeptidyl peptidase 4 (DPP4) inhibitors which in the Investigator's opinion could interfere with glucose or lipid metabolism 90 days prior to screening
7. Cancer (except basal cell skin cancer or squamous cell skin cancer) or any other clinically significant disorder, except for conditions associated with type 2 diabetes history, which in the investigators opinion could interfere with the results of the trial
8. Inflammatory bowel disease
9. Cardiac disease defined as: Decompensated heart failure (NYHA class III-IV) and/or diagnosis of unstable angina pectoris and/or myocardial infarction within the last 6 months
10. Previous bowel resection
11. Body mass index <18.5 kg/m2
12. Females of childbearing potential who are pregnant, breast-feeding, intend to become pregnant or are not using adequate contraceptive methods
13. Clinical signs of diabetic gastroparesis
14. Impaired liver function (transaminases > two times upper reference levels)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2012-08; Primary Completion 2013-07 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Change in ambulatory blood pressure | 50 days
  Change in 24h BP from day 1 to day 49 (baseline to end of treatment) and time to statistically significant change in BP 24h after initiation of or increased dose of liraglutide

SECONDARY OUTCOMES:
Change in ECV | 50 days
  Changes in ECV (measured by GFR), urinary sodium, weight, arterial stiffness and daily home-BP, from day 1 to day 49 (baseline to end of treatment).
Washout analysis | 21
  Change in 24h BP, ECV, weight, arterial stiffness from day 49 to day 70th

CONTACTS AND LOCATIONS:
Overall Officials: Peter Rossing, MD, Principal Investigator — Steno Diabetes Centes
Locations (1):
- Steno Diabetes Center, Gentofte Municipality, Denmark

REFERENCES:
- [Derived] von Scholten BJ, Hansen TW, Goetze JP, Persson F, Rossing P. Glucagon-like peptide 1 receptor agonist (GLP-1 RA): long-term effect on kidney function in patients with type 2 diabetes. J Diabetes Complications. 2015 Jul;29(5):670-4. doi: 10.1016/j.jdiacomp.2015.04.004. Epub 2015 Apr 11. PMID 25935863